CLINICAL TRIAL: NCT06611787
Title: A Comprehensive Registry Study of the Whole Life Cycle of Patients With Congenital Heart Diseases
Brief Title: A Comprehensive Registry Study of the Whole Life Cycle of Patients With CHD
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 2024 No. (1) RSTE
Record Dates: First submitted 2024-08-15; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Discarded myocardial samples removed during surgery, and blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to collect data on the prevalence, intervention, and prognosis of congenital heart disease (CHD) in Chinese patients across their entire lifecycle. From the diagnosis of CHD in fetuses, to early treatment of severe CHD in neonates, to standardized perinatal diagnosis and treatment of CHD patients with concurrent pregnancy, the study employs a cyclical model consisting of evaluation, training, improvement, and re-evaluation. The goal is to enhance the diagnostic and treatment capabilities of participating hospitals, especially for complex CHD cases, and promote standardized clinical practices in cardiovascular disease treatment among these hospitals. This will ultimately improve the quality of medical services provided to cardiovascular patients and serve as a basis for exploring CHD treatment guidelines suitable for China.

The project will be implemented by Capital Medical University Affiliated Beijing Anzhen Hospital and the National Clinical Research Center for Cardiovascular Diseases. The plan is to involve more than 20 hospitals over the next five years. An independent website will be created for data collection, education and training, as well as experience sharing among participating hospitals. Starting from January 1, 2024, each hospital will continuously collect CHD inpatient cases on a monthly basis. The project team will regularly analyze and report on the completion of key medical quality evaluation indicators for each hospital. They will provide guidance measures such as education, training, experience sharing, and on-site investigations to address identified issues, helping hospitals improve medical quality. Hospitals that demonstrate excellence and significant improvement will be recognized and commended, driving overall improvement in the quality of cardiovascular medical care in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients with various congenital heart diseases

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with various congenital heart diseases.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
The mortality of the first week after surgery | Duration of hospital stay (an expected average of 1 week)
  Intraoperative surgeries encompass a broad range of procedures performed during a surgical operation, often involving complex and high-risk interventions. In terms of in-hospital mortality within 1 weeks after surgery, the risk associated with intraoperative surgeries can be elevated due to factors, the complexity of the procedure, and potential complications.
  Routine neonatal surgeries, on the other hand, are procedures commonly performed on newborns, often to address congenital anomalies or other medical conditions present at birth. While these surgeries are generally considered safer than more complex intraoperative procedures, there is still a risk of in-hospital mortality within 1 week after surgery, particularly for neonates with pre-existing health issues or complications during the surgical process. Close monitoring and prompt intervention are crucial to minimize this risk and ensure the best possible outcomes for neonatal patients

SECONDARY OUTCOMES:
The ratio of newborns receiving integrated prenatal and postnatal diagnosis and treatment; | Duration of hospital stay (an expected average of 1 week) and 5 years after discharge
The ratio of intraoperative surgeries among all neonatal surgeries; | Duration of hospital stay (an expected average of 1 week) and 5 years after discharge
The rate of Medium- and long-term survival rates, and re-operations | Duration of hospital stay (an expected average of 1 week) and 5 years after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing AnZhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No